CLINICAL TRIAL: NCT05879237
Title: Role of Vitamin D Supplementation as an Adjuvant Therapy inTreatment of Helicobacter Pylori in Children
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Minia University (Other)
Collaborators: Ain Shams University (Other)
Responsible Party: Principal Investigator, Shimaa Mohamed Yassin, Doctor, Minia University
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2021:42
Record Dates: First submitted 2023-05-18; First posted 2023-05-30 (Actual); Last update posted 2023-05-30 (Actual); Status verified 2023-05

CONDITIONS: Helicobacter Pylori Infection
MeSH Terms: interventions — Cholecalciferol

STUDY DESIGN:
Intervention Model Description: To study the efficacy of vitamin D in conjunction with Helicobacter pylori treatment in children in eradication of helicobacter pylori.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Triple therapy therapy and vitamin D3 (Active Comparator): Vitamin D3 ,1000 unit ,once daily, oral, for 1 month plus the standard triple therapy of H pylori (double antibiotics and proton pump inhibitor)
  Interventions: Drug: Vitamin D3; Drug: Helicobacter pylori triple therapy
- Triple therapy only (Active Comparator): Standard triple therapy of H pylori
  Interventions: Drug: Helicobacter pylori triple therapy

INTERVENTIONS:
Drug: Vitamin D3 — Vitamin D3 ,1000 unit ,once daily, oral, for 1 month plus triple therapy
  Other Names: cholecalciferol
  Arms: Triple therapy therapy and vitamin D3
Drug: Helicobacter pylori triple therapy — Triple therapy which is: amoxcillin on 50 mg/kg/day for 2 weeks, Clarithromycin 20mg/kg/day for 2 weeks and proton pump inhibitor
  3.ppi 1mg/kg/day for 1month

SUMMARY:
To study the efficacy of vitamin D in conjunction with Helicobacter pylori treatment in children in eradication of helicobacter pylori.

DETAILED DESCRIPTION:
o study the efficacy of vitamin D in conjunction with Helicobacter pylori treatment in children in eradication of helicobacter pylori.

our study include 2 patient groups:

1. st group included 100 child diagnosed Helicobacter pylori infection by upper gastrointestinal endoscopy and biopsies with pathology, will receive H.pylori eradication treatment and vitamin D as an adjuvant therapy .
2. nd group will also diagnosed Helicobacter pylori infection by upper gastrointestinal endoscopy and biopsies with pathology, will receive H.pylori eradication treatment only.

Helicobacter pylori treatment :

1. amoxcillin on 50 mg/kg/day for 2 weeks
2. clarithromycin 20mg/kg/day for 2 weeks
3. proton pump inhibitor 1mg/kg/day for 1month Vitamin d dose..1000unit /day for 1 month

ELIGIBILITY:
Inclusion Criteria:

- Age:4-18 years children with symptomatic H pylori infection presenting with (epigastric pain, persistent vomiting and hematemesis)diagnosed by upper gastrodeudonoscopy , rapid urease test and histopathologic examination of gastric biopsies from antrum and body of the stomach.

Exclusion Criteria:

* Patient on vitamine D supplémentation
* Patient who has defect in vitamin D metabolism (chronic renal and hepatic patients, malabsorption syndromes)
* Patients who had received treatment of H.pylori previously .

Ages: 4 Years to 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200 (Estimated)
Dates: Start 2023-06-01 (Estimated); Primary Completion 2023-12-01 (Estimated); Study Completion 2023-12-10 (Estimated)

PRIMARY OUTCOMES:
Role of Vitamin D Supplementation as an Adjuvant Therapy inTreatment of Helicobacter Pylori in Children | Six month
  eradication of h pylori in children

CONTACTS AND LOCATIONS:
Overall Officials: samir M mounir, ass prof, Study Director — Minia University, faculty of medicine; Yosra M awad, lecturer, Study Director — ain shams university .faculty of medicine; shimaa M yassin, ass lect, Principal Investigator — Minia University, faculty of medicine

IPD SHARING:
Plan to Share IPD: Yes
study role of vitamin D supplementation as an Adjuvant Therapy IN Treatment of Helicobacter Pylori in Children
Supporting Information: Study Protocol, SAP, ICF, CSR, Analytic Code
Time Frame: 6 month
Access Criteria: study role of vitamin D supplementation as an Adjuvant Therapy IN Treatment of Helicobacter Pylori in Children revised by dr yosra m awad
URL: http://Yosraawad@med.asu.edu.eg